CLINICAL TRIAL: NCT00205127
Title: Comparison of Cardiac Perfusion by O15-water and F17-fluoromethane PET
Brief Title: Cardiac Water and Fluoromethane Cardiac PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003-241
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Volunteers
Keywords: Cardiac PET imaging; Radiopharmaceutical tracers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac PET imaging- rest and pharmacological stress

SUMMARY:
In this study we are looking at the blood flow to the heart using two different chemical tags or tracers that give off a low level of radiation. The tracers used in this study are called O15-water and F17-fluoromethane. These tracers mix with the blood and will move through the body. The researchers will use positron emission tomography (PET scans)to track the tracers as they moe through the heart and chest.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 40 years old 2. Willing to provide written informed consent

Exclusion Criteria:

* 1. A history of CAD 2. A history of active bronchospasm or asthma on theophylline bronchodilators 3. A history of any cardiac risk factors including: HTN, Diabetes, Hyperlipidemia, Smoking, and premature CAD in immediate family member 4. A history of liver disease or other significant disease 5. Females who are pregnant or lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2004-01; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
-- implement myocardial perfusion quantification for O15-labeled water at rest and with pharmacologic stress, | assess at time of PET scan
-- determine the biodistribution of fluoromethane in the thorax to see if it is usable for a cardiac perfusion tracer, | assess at time of PET Scan

SECONDARY OUTCOMES:
--develop initial methods for quantification of myocardial perfusion if applicable for labeled fluoromethane. | assess at time of PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Charles K Stone, MD, Principal Investigator — Univeristy of Wisconsin
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States